CLINICAL TRIAL: NCT04110561
Title: Evaluation of Safety and Performance of the Atalante System With Patients With Lower Limb Paralysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wandercraft (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TPL005
Record Dates: First submitted 2019-09-26; First posted 2019-10-01 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Spinal Cord Injuries; Paraplegia; Paralysis, Lower Limbs; Lower Extremity; Robotics
Keywords: Spinal Cord Injuries; Paraplegia; Paralysis, Lower Limbs; Lower Extremity; Robotics; Physiotherapy; Rehabilitation; Powered Exoskeleton; Walking; Ambulation
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spinal Cord Injury patients with motor complete paralysis (Other)
  Interventions: Device: Use of the Atalante exoskeleton

INTERVENTIONS:
Device: Use of the Atalante exoskeleton — A session basically includes a stand up, walks over a distance of 10 meters, exercises, U-turns and a sitting

SUMMARY:
The study is a prospective, open, bicentric and observational study. It is conducted to assess the safety and performance of the Atalante exoskeleton system with patients with lower limb paralysis.

The principal objective is to assess the performance of the Atalante system in performing ambulatory functions with motor complete SCI patients characterized by the success rate in performing a 10mWT at the last session of training with the Atalante system.

ELIGIBILITY:
Inclusion Criteria:

* Motor complete traumatic Spinal Cord Injury (AIS A and B) since at least 4 months
* Spinal Injury Level between AIS T5 and AIS T12
* Able to verticalize on a daily basis
* Height: between approximately 1.60 and 1.90 m. More specifically, Atalante is able to accommodate the following limb lengths:

  * Thigh: 380-460 mm
  * Distance between the ground and the joint space of the knee (to be measured while wearing the shoes they intend to wear with Atalante):

    * 457-607 mm for patient with an ankle dorsiflexion ≥ 16°
    * 457-577 mm for patient with an ankle dorsiflexion between 13° et 16°
    * 457-567 mm for patient with an ankle dorsiflexion between 10° et 13°
    * 457-557 mm for patient with an ankle dorsiflexion between 0° et 10° o Hip width less of equal to 460 mm when seated
* Maximum weight: 90 kg
* Patient having given his written consent

Exclusion Criteria:

* Patients whose joint centers cannot be aligned Atalante's
* Ranges of motion below:

  * Hip: 115° flexion, 15° extension, 17° abduction, 10° adduction, 10° medial rotation, 20° lateral rotation
  * Knee: 5° extension, 110° flexion
  * Ankle: 0° dorsiflexion, 9° plantar flexion, 18° inversion and eversion
* Severe spasticity (greater than 3 on the modified Ashworth scale) of the adductor muscles, hamstrings, quadriceps and triceps surae
* Pregnant or lactating woman
* Unbalanced psychiatric or cognitive status which may interfere with an appropriate use of the device
* Other neurological disorder
* History of osteoporotic fracture and/or disease or treatment responsible for a secondary osteoporosis
* Active implantable medical device
* Evolutive intercurrent disease: pressure sore, infection, venous thrombosis
* Unstable and unhealed limb and pelvic fracture
* Unstable spine
* Severe illness which may interfere with the verticalized posture and tolerance to effort
* Evolutive osteoma
* Syringomyelia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-05 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the clinical investigation is defined by the success or failure at the 10 Meter Walk Test (10mWT) at the latest session. | At study completion, up to 3 weeks
  The 10mWT is used to assess walking speed in meters/second (m/s) over a short distance.
  A clear pathway of at least 10-meter length is drawn. The start and the end point of a 10-m walkway is marked by lines.
  The patient starts a few steps prior the starting line; during the few steps needed to reach the starting line, the physiotherapist should stabilize the exoskeleton in the frontal plane. When the patient's first foot crosses the starting line, the test begins, and the stopwatch is started. The stopwatch is stopped at the end of the 10 meters in case of success, that is to say when the patient crosses the end line.
  The total time taken to ambulate is recorded. The distance covered is then divided by the total time (in seconds) taken to ambulate and recorded in meters per seconds.
  In case of failure, the distance walked by the patient is measured and recorded, and the speed to walk this distance is calculated as described above.

SECONDARY OUTCOMES:
Capacity of patient in walking defined by Success / Failure on a 10mWT test at the 6th session. | At study mid-term, 10 days in average
The maximum distance walked during the 10mWT at the 6th and 12th sessions. | At study mid-term, 10 days in average and at study completion, up to 3 weeks
The average walking speeds during the 10mWT at the 6th and 12th sessions. | At study mid-term, 10 days in average and at study completion, up to 3 weeks
Capacity of the patient to perform verticalization as defined by the test "Stand-up" at the 6th and 12th sessions. | At study mid-term, 10 days in average and at study completion, up to 3 weeks
Capacity of a standing patient to reach a sitting position as defined by the test "Sit down" at the 6th and 12th sessions. | At study mid-term, 10 days in average and at study completion, up to 3 weeks
Ability of the patient to maintain a stand still position for 2 minutes as defined by the test "Stand without support for 2 minutes" at the 6th and 12th sessions. | At study mid-term, 10 days in average and at study completion, up to 3 weeks
Ability of the patient to lean with extended arm in a standing position (90° arms) at the 6th and 12th sessions. | At study mid-term, 10 days in average and at study completion, up to 3 weeks
Ability of the patient to perform a U-turn in less than 3 minutes as defined by the test "Make a U-turn" at the 6th and 12th sessions. | At study mid-term, 10 days in average and at study completion, up to 3 weeks
Average scores on Borg CR-10 simple perception scale for the perceived exertion at the 6th and 12th sessions. | At study mid-term, 10 days in average and at study completion, up to 3 weeks
  Rating of perceived exertion (RPE) is a widely used and reliable indicator to monitor and guide exercise intensity.
  The scale allows individuals to subjectively rate their level of exertion during exercise or exercise testing.
  Developed by Gunnar Borg, it is often also referred to as the Borg Scale. Despite being a subjective measure of exercise intensity, RPE scales provide valuable information when used correctly.
  The revised category-ratio scale (0 to 10 scale) is used:
  * 0 Null
  * 1 Very easy
  * 2 Somewhat easy
  * 3 Moderate
  * 4 Somewhat hard
  * 5 Hard
  * 6
  * 7 Very hard
  * 8
  * 9
  * 10 Very, very hard
Average scores of safety perceived by the patient on a 7-point Likert scale 7 levels at the 6th and 12th sessions. | At study mid-term, 10 days in average and at study completion, up to 3 weeks
  A Likert scale is a psychometric scale commonly involved in research based on survey questionnaires. Here, the respondents specify their level of agreement or disagreement using a symmetric agree-disagree scale for a series of statements while responding to a particular Likert questionnaire item. The range of Likert scale captures the intensity of their feelings for a given item.
  The Likert scale ratings are:
  1. Strongly disagree
  2. Disagree
  3. Disagree somewhat
  4. Neither agree nor disagree
  5. Agree somewhat
  6. Agree
  7. Strongly agree
  The perceived safety is evaluated with the 7-point Likert scale on the following statement:
  "I felt safe during the test"
Observation of the skin condition was made before and after each session on the subject's back, thighs, knees and feet. | Throughout study completion, an average of 3 weeks
Comparison of the NBD score before the 1st session and after the 12th session. | At study start, day 1 and at study completion, up to 3 weeks
  The neurogenic bowel dysfunction score is a questionnaire including questions about background parameters, faecal incontinence, constipation, obstructed defecation, and impact on quality of life. The NBD score is constructed from items with acceptable reproducibility and validity that were significantly associated with impact on quality of life. The type of the stool depends on the time it spends in the colon.
Comparison of the Bristol scale before the 1st session and after the 12th session. | At study start, day 1 and at study completion, up to 3 weeks
  The Bristol Stool Chart is:
  * Type 1: Separate hard lumps, like nuts (hard to pass);
  * Type 2: Sausage-shaped but lumpy;
  * Type 3: Like a sausage but with cracks on its surface;
  * Type 4: Like a sausage or snake, smooth and soft;
  * Type 5: Soft blobs with clear-cut edges (passed easily);
  * Type 6: Fluffy pieces with ragged edges, a mushy stool;
  * Type 7: Watery, no solid pieces. Entirety liquid.
  Type 1, 2 and 3 indicate constipation. Type 4 and 5 are ideal stools. Type 6 and 7 indicate diarrhea and urgency.
Definition of the voiding mode at the 1st and 12th sessions. | At study start, day 1 and at study completion, up to 3 weeks
  The management of neurogenic bladder dysfunction is crucial in the management of paraplegic patients as it affects the morbidity of these patients. The voiding mode is described. The self-survey is the standard treatment when the subject has an overactive bladder. The mictionnel mode will be informed before the first session, and at the end of the last session with the exoskeleton using an ISCOS questionnaire (International Spinal Cord Society questionnaire).
Qualiveen score at the 1st and 12th sessions. | At study start, day 1 and at study completion, up to 3 weeks
  The Qualiveen score is developed as a condition-specific quality of life measurement for individuals with SCI who have urinary disorders. It contains 4 domains:
  * Limitation/ Inconvenience;
  * Constrains/ Restrictions;
  * Fears;
  * Feelings/ Impact on Daily Life.
  The test-retest reliability is high6.
Spasticity according to the Modified Ashworth scale at the 1st and 12th sessions. | At study start, day 1 and at study completion, up to 3 weeks
  The Modified Ashworth Scale measures spasticity in patients with lesion of the Central Nervous System. The relationship between the raters' judgments was significant and the reliability was good. (PMID: 3809245)
  The scoring is:
  * 0: No increase in muscle tone
  * 1: Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  * 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  * 2: More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  * 3: Considerable increase in muscle tone, passive movement difficult
  * 4: Affected part(s) rigid in flexion or extension
  Muscles evaluated are adductor, hamstring, triceps sural and quadriceps.
Heart rate measurement at rest and after the 10mWT at the 1st, 6th and 12th sessions. | At study start, day 1, at study mid-term, 10 days and at study completion, up to 3 weeks
Comparison of the Visual Analogue Pain Scale at the 1st and 12th sessions. | At study start, day 1 and at study completion, up to 3 weeks
  The Numeric Pain Rating Scale measures the subjective intensity of pain. The NPRS is an 11-points scale from 0 to 10: "0" = no pain; "10" = the most intense pain imaginable.
  The subject is asked to make pain rating corresponding to the current pain experienced.
Comparison of the NPSI scores at the 1st and 12th sessions. | At study start, day 1 and at study completion, up to 3 weeks
  NPSI (Neuropathic Pain Sumptom Inventory) renders it suitable for the evaluation of the different dimensions of neuropathic pain syndromes. The reliability of the different descriptors appears to be sufficient.
  It allows to quantify the various pain symptoms that can be grouped into five dimensions (burn, deep pain, paroxysmal pain, pain caused, paresthesia / dysesthesia)
Patient Global Impression of Improvement (PGI-I) at the 12th session. | At study completion, up to 3 weeks
  The Patient Global Impression of Improvement (PGI-I) is a global index that may be used to rate the response of the use of Atalante on the bowel function.
  The subject should check the number that best describes how the twelfth session condition is, compared with how it has been at the first session for the bowel function:
  1. Very much better
  2. Much better
  3. A little better
  4. No change
  5. A little worse
  6. Much worse
  7. Very much worse
Average scores of the 7-point Likert scale for ergonomics at the 12th session. | At study completion, up to 3 weeks
  At the end of the twelfth session, the patient evaluates the interfaces and the ergonomics of Atalante (shape of the remote, mode, symbol) and the perceived safety and the level of assistance during transfer from the wheelchair to Atalante with a Likert scale.
  The Likert scale is a questionnaire where the subject chooses among seven-point scales:
  1. Strongly disagree
  2. Disagree
  3. Disagree somewhat
  4. Neither agree nor disagree
  5. Agree somewhat
  6. Agree
  7. Strongly agree
Time of installation of the patient in the exoskeleton at the 12th session. | At study completion, up to 3 weeks
Assistance level for each fastener at the 12th session. | At study completion, up to 3 weeks
  The level of assistance is specified for each attachment (thigh, knee and foot straps). The levels of assistance are:
  * Without assistance;
  * With the assistance of one health professional;
  * With the assistance of two health professional.
Average scores of the 7-point Likert scale for exoskeleton attachment questionnaire at the 12th session. | At study completion, up to 3 weeks
  At the end of the twelfth session, the strapping system is evaluated using a 7-point Likert scale:
  1. Strongly disagree
  2. Disagree
  3. Disagree somewhat
  4. Neither agree nor disagree
  5. Agree somewhat
  6. Agree
  7. Strongly agree
Evaluation of sitting balance using the Boubee test at the 1st and 12th sessions. | At study start, day 1 and at study completion, up to 3 weeks
  This test evaluates the ability of the subject to balance in sitting position during disturbances induced by movements of the upper limbs. The subject is sitting without back's support and with both feet on the ground. The subject is asked to do six tasks from the easiest to the hardest. The subject must pass the task to test the next task. The score is defined by the last passed task. The sitting balance is evaluated at the first and at the last session.
Adverse events collection at each session. | Throughout study completion, an average of 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Kerdraon, Dr, Principal Investigator — Centre mutualiste de Rééducation et de Réadaptation de Kerpape
Locations (2):
- France (2):
  - Centre Jacques Calvé - Fondation Hopale, Berck
  - Centre mutualiste de Rééducation et de Réadaptation de Kerpape, Ploemeur

IPD SHARING:
Plan to Share IPD: No